CLINICAL TRIAL: NCT00440388
Title: An Open-label, Multicenter, Phase II Study of AT-101 in Combination With Rituximab in Patients With Untreated, Grade I-II, Follicular Non-Hodgkin's Lymphoma
Brief Title: Safety & Efficacy Study of AT-101 in Combination w/ Rituximab in Previously Untreated Grade I-II Follicular Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascenta Therapeutics (Industry)
Responsible Party: Jeffrey Brill, Associate Director, Clinical Development, Ascenta Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-101-CS-203
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Follicular Lymphoma
Keywords: cancer; lymphoma; Non-Hodgkin's; Non-Hodgkins; AT-101; AT101; Rituxan; Rituximab
MeSH Terms: conditions — Lymphoma, Follicular; Neoplasms; Lymphoma | interventions — gossypol acetic acid; Rituximab

INTERVENTIONS:
Drug: AT-101 — AT-101 30 mg orally for 21 of 56 days, every cycle. Cycle = 56 days; Max of 5 cycles.
Drug: Rituximab — Rituximab 375mg/m2 IV once per week for four weeks during 1st cycle, 375mg/m2 IV once per cycle for cycles 2-5. Cycle = 56 days; Max of 5 cycles.

SUMMARY:
This is a phase II clinical trial in patients who have not received systemic treatment for follicular non-Hodgkin's lymphoma. The study combines rituximab, an approved drug for this disease, with AT-101, an experimental drug. The hypothesis is that by adding AT-101 to the rituximab regimen, improvement to patients' response to the treatment will be observed verses rituximab alone.

DETAILED DESCRIPTION:
Further Study Details provided by Ascenta.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, previously untreated Grade I-II follicular B-cell non-Hodgkin's lymphoma (stage I, II, III and IV). Patients may have received radiation therapy to one lymph node region; Stage I or II patients must have relapsed after prior radiation therapy to be eligible;
* Patients with any FLIPI score may participate. Patients with FLIPI scores 3-5 may be enrolled with asymptomatic disease, or without worsening disease or disease related-symptoms; however patients with FLIPI scores of 0-2 must have evidence of worsening disease;
* ECOG performance status 0-1;
* Measurable disease;
* Adequate hematological function as indicated by:

  * Absolute neutrophil count (ANC) >1,000/µL; +Hemoglobin >8 g/dL (It is acceptable to transfuse PRBC to achieve this criterion);
  * Platelet count >50 x 109/L.
* Adequate hepatic and renal function as indicated by:

  * Serum creatinine ≤2.0 mg/dL;
  * Serum albumin ≥2.5 g/dL;
  * Total bilirubin ≤1.5 x upper limit of normal (ULN);
  * Serum AST and ALT ≤1.5 x ULN.
* Able to swallow and retain oral medication

Exclusion Criteria:

* Patients who have severe lymphoma-related symptoms requiring a rapid response to therapy (e.g., requirement for cytoreduction due to advanced disease or organ compromise, respiratory compromise because of large effusions or airway obstruction, bowel obstruction, ureteral obstruction, and chylous ascites);
* Active symptomatic fungal, bacterial and/or viral infection including, but not limited to active HIV or viral hepatitis (A, B or C);
* History of hepatitis B infection;
* Any B-cell, T-cell or transformed lymphoma other than histologically confirmed follicular non-Hodgkin's lymphoma;
* Central nervous system (CNS) lymphoma, CNS or leptomeningeal involvement by lymphoma (treated or in remission), HIV-related lymphoma, or patients with symptoms suggesting HIV infection;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
complete or partial remission of disease | 8 weeks

SECONDARY OUTCOMES:
duration of complete or partial remission of disease | 10 months
number of participants with adverse events | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Ascenta Therapeutics, Inc.
Locations (28):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Rocky Mountain Cancer Center-Aurora, Aurora, Colorado
  - Florida Cancer Institute, Hudson, Florida
  - Florida Cancer Institute, New Port Richey, Florida
  - Cancer Care & Hematology Specialists of Chicagoland, Arlington Heights, Illinois
  - Central Indiana Cancer Centers, Fishers, Indiana
  - University of Michigan Cancer Center, Ann Arbor, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Hematology/Oncology Associates, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - Duke University Medical Center, Durham, North Carolina
  - Northwest Cancer Specialists, Portland, Oregon
  - The Jones Clinic, Germantown, Tennessee
  - Texas Oncology, P.A., Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - Allison Cancer Center, Midland, Texas
  - HOAST - New Braunfels, New Braunfels, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Hematology Oncology Physicians of Texas, Richardson, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Virginia Oncology Associates, Chesapeake, Virginia
  - Oncology and Hematology Associates of SW Virginia, Inc., Salem, Virginia
  - Cancer Care Northwest, Spokane, Washington
  - St. Mary's Medical Center, Huntington, West Virginia